CLINICAL TRIAL: NCT02701608
Title: Oral Switch During Treatment of Left-sided Endocarditis Due to Multi-susceptible Staphylococcus (Relais Oral Dans le Traitement Des Endocardites à Staphylocoques Multi-sensibles)
Brief Title: Oral Switch During Treatment of Left-sided Endocarditis Due to Multi-susceptible Staphylococcus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RODEO 1
Record Dates: First submitted 2016-01-28; First posted 2016-03-08 (Estimated); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Infective Endocarditis
MeSH Terms: conditions — Endocarditis | interventions — Levofloxacin; Fluoroquinolones; Rifampin; Oxacillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral switch treatment (Experimental): Oral switch to the combination of levofloxacin and rifampicin
  Interventions: Drug: Levofloxacin; Drug: Rifampicin
- Conventional IV treatment according to european guidelines (Active Comparator): Conventional IV treatment of staphylococci IE (European guidelines 2015)
  Interventions: Procedure: Conventional IV treatment of staphylococci IE following European guidelines 2015 including cloxacilline, oxacilline,gentamicine,vancomycine,rifampicine

INTERVENTIONS:
Drug: Levofloxacin — levofloxacin 500 mg x1/day (for patients ≤70kg) or levofloxacin 750 mg x1/day (for patients >70kg)
  Other Names: Fluoroquinolones
  Arms: Oral switch treatment
Drug: Rifampicin — rifampicin 600mg x1/day (for patients ≤70kg) or rifampicin 900mg x1/day (for patients >70kg)
  Arms: Oral switch treatment
Procedure: Conventional IV treatment of staphylococci IE following European guidelines 2015 including cloxacilline, oxacilline,gentamicine,vancomycine,rifampicine — Conventional IV treatment of staphylococci IE following European guidelines 2015 including cloxacilline, oxacilline,gentamicine,vancomycine,rifampicine
  Arms: Conventional IV treatment according to european guidelines

SUMMARY:
Infective endocarditis (IE) is a serious infection with a significant burden for patients and hospitals (in France, median length of hospital stay = 43 days), partly due to the long duration of intravenous (IV) antibacterial treatment recommended by international guidelines, between 4 and 6 weeks in most situations.

A recent survey of practices regarding the management of IE in France showed that a switch from IV to oral antibiotics is feasible, when patients with left-sided Staphylococcus IE are stable after an initial course of IV antibiotic treatment, with or without valvular surgery.

These practices have not been associated with unfavourable outcome, while significantly reducing the duration and cost of hospitalization, the risk of nosocomial infection, and patients' discomfort.

There has been no randomized controlled trial (RCT) in the field of IE over the last 20 years; current guidelines are mostly based on expert advice, in vitro studies, animal experiments, or clinical studies performed before the 90's.

The RODEO 1 project is an unprecedented opportunity to bring back evidence-based medicine in the field of IE.

Most experts acknowledge that the pharmacological PK/PD characteristics of antibiotics such as fluoroquinolones and rifampicin allow a high level of efficacy in the treatment of IE when orally administrated after an IV period of induction.

It's needed to conduct RCTs that clearly demonstrate the clinical non-inferiority of this strategy for multisusceptible staphylococci with a benefit regarding costs.

The RODEO 1 project corresponds to one pragmatic trial assessing the impact of a switch strategy, making it a comparative effectiveness trial that should be able to feed the next revision of IE international guidelines and to change practices in IE management.

DETAILED DESCRIPTION:
The RODEO 1 study is designed to determine the safety and efficacy of partial oral treatment of IE compared with traditional full-length parenteral treatment. Our primary objective is to demonstrate that in patients with left-sided multi-susceptible Staphylococcus who have received at least 10 days of IV antibiotic treatment with or without valvular surgery, a switch to an oral combination of rifampicin and fluoroquinolones between Day 10 and Day 28 after initiation of the IV antibiotic treatment, is not inferior to the continuation of the conventional IV antibiotic treatment regarding to treatment failure within 3 months after the end of antibiotic treatment.

Nationwide, noninferiority, multicenter, randomized, controlled, open-label trials.

Randomisation will only be offered to patients who have received at least 10 days of IV conventional antibiotic treatment of IE, and fulfil the inclusion criteria.

Randomisation will take place between Day 10 and Day 28 after initiation of parenteral antibiotic therapy or valvular surgery, thus ensuring to have at least 14 days of oral therapy in the experimental group.

Patients will be eligible whether they have undergone valvular surgery or not. This will imply that surgery procedure prior to randomisation will be heterogeneous, but randomisation will be stratified on the requirement of valvular surgery as part of the treatment of the current episode of IE or not.

ELIGIBILITY:
Inclusion Criteria:

* Left-sided IE (Defined according to Duke criteria) on native or prosthetic valve
* due to one isolate of Staphylococcus sp. (S. aureus or coagulase negative staphylococci, CNS) susceptible to levofloxacin and rifampicin
* in an adult ≥18 year old
* appropriate parenteral antibiotics treatment received for at least 10 days
* in case of valvular surgery, appropriate parenteral antibiotics treatment received for at least 10 days after valvular surgery
* planned duration of antibiotics will extend for at least 14 days at the time of randomisation i.e. a potential switch to oral treatment between Day 10 and Day 28 thus ensuring to have at least 14 days of oral therapy remaining in the experimental group
* apyrexia (temperature < 38°C) at each time point during the last 48 hours (at least two measures/day) at the time of randomisation
* blood cultures have been sterile for at least 5 days at the time of randomisation
* informed, written consent obtained from patient
* subject covered by or having the rights to French social security

Exclusion Criteria:

* body mass index <15 kg/m² or > 40 kg/m²
* glomerular filtration rate < 50 ml/min/1,73m²
* patient unable or unwilling to take oral treatment (digestive intolerance, significant malabsorption) at the time of randomisation
* expected difficulties regarding compliance with oral antibiotic treatment or follow-up (e.g. severe cognitive impairment, severe psychiatric disease...)
* patient without entourage to support and watch him at discharge
* valvular surgery planned within the next 6 months
* patients with cardiac devices (pace-maker, implantable cardiac defibrillator) and suspected device-related IE (vegetation on the leads) if removal of the device was not performed
* breast feeding or pregnant women, or women on childbearing age without effective contraception
* expected duration of follow-up < 7 months at the time of randomisation (e.g. expected life expectancy < 7 months, patient living abroad...)
* past medical history of IE in the last 3 months
* other infection requiring parenteral antibiotic therapy
* taking of an estrogen-progesterone treatment interacting with rifampicin
* patient with contra-indication to oral antibiotics administered in the experimental arm (i.e. fluoroquinolones or rifampicin ) - including anticipated non-manageable drug interactions with rifampicin, and allergy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2016-02-29 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
Treatment failure | up to 3 months after the end of antibiotic treatment
  Failure is a composite outcome defined by death from all causes and/or symptomatic embolic events and/or unplanned valvular surgery and/or a microbiological relapse (with the primary pathogen).

SECONDARY OUTCOMES:
death from all-cause | up to 6 months after the end of antibiotic treatment
  death from all-cause
number of symptomatic embolic events | up to 6 months after the end of antibiotic treatment
  secondary osteo-articular, splenic or brain localization
unplanned valvular surgery | up to 6 months after the end of antibiotic treatment
  unplanned valvular surgery
relapse of positive blood cultures | up to 6 months after the end of antibiotic treatment
  relapse of positive blood cultures with the primary pathogen
microbiological relapse with a different pathogen from the primary pathogen | up to 6 months after the end of antibiotic treatment
  Relapse of positive blood cultures with a different pathogen within 3 months after the end of antibiotic therapy
Echocardiography | up to 6 months after the end of antibiotic treatment
  An apparition, an increase or decrease of the following items: vegetation, abscess, perforation, fistula, dehiscence of a prosthetic valve, will be searched at each ultrasound examination at : the end of antibiotic treatment, at 3 months and 6 months after the end of antibiotic treatment
Catheter related adverse events | up to 6 months after the end of antibiotic treatment
  Catheter-related AE: infectious (e.g. catheter-related bacteraemia) or non-infectious catheter-related complications (e.g. extravasation).
other healthcare-acquired infections | up to 6 months after the end of antibiotic treatment
  other healthcare-acquired infections, including urinary tract infections, pneumonia, surgical site infection, Clostridium difficile infections
Number of participants with an antibiotic modification | up to the end of antibiotic treatment
  All change regarding antibiotic treatment administered will be recorded (drug, dose or duration)
Quality of life | up to 6 months after the end of antibiotic treatment
  An assessment of patient's quality of life will be done at the end of antibiotic treatment, at 3 months and 6 months after the end of antibiotic treatment, using the EuroQol Five Dimensions (EQ5D3L)
number of participants with a switch back from oral to IV antibiotic treatment | up to the end of antibiotic treatment
  For experimental group only . An assessment of the need for a return to parenteral antibiotic in the experimental group.
Compliance with oral antibiotic treatment | up to 4 weeks after randomisation
  For experimental group only. The assessment of compliance with oral antibiotic treatment will be carried out at each visit during the treatment period.
Cost per patient | up to 6 months after the end of antibiotic treatment
  Analysis using data from three centers (Tours, Rennes, Nancy) to compare both strategy (oral switch vs. pan-IV) for the cost per patient
Budget impact analysis (BIA) | up to 6 months after the end of antibiotic treatment
  With data from three centers (Tours, Nancy, Rennes). With data from three centers (Tours, Nancy, Rennes). Allow to estimate the financial consequences of the adoption and diffusion of a new health intervention (the oral strategy). BIA must be calculated on a yearly basis.
Utility score and incremental cost-utility ratio (ICUR) | up to 6 months after the end of antibiotic treatment
  With data from all centers. An assessment of the health related quality of life of the patient will be carried out using a simple generic questionnaire, the EuroQol Five Dimensions (EQ5D3L), recommended by the Washington Panel on Cost Effectiveness (utility) in Health and Medicine, with a cardinal scale and validated French version (http://www.euroqol.org)Quality of life will be assessed 4 times: at baseline, at the end of antibiotic treatment, at 3 months after end of antibiotic treatment and at the final visit.
Length of hospital stay | up to 6 months after the end of antibiotic treatment
  With data from all centers. Length of hospital stay will be calculated as duration between day of start of hospitalization and day of discharge (distinguishing rehabilitation care unit). In case a patient dies during hospitalization, death will be considered as a competing event to discharge.
Residual concentration of antibiotics | 7 days
  Pharmacokinetic analysis for the experimental group only: residual concentrations of levofloxacin and rifampicin, or amoxicillin, after 7 days of oral treatment (i.e. at visit 2).
Biological collection for further analysis on endocarditis | up to 6 months after the end of antibiotic treatment
  A biological collection will be constituted in order to perform further biological and genetic analysis of endocarditis (i.e. inflammatory markers of efficacy and genetic markers that predispose to endocarditis).

CONTACTS AND LOCATIONS:
Overall Officials: Louis BERNARD, MD,PHD, Principal Investigator — CHRU TOURS
Locations (45):
- France (45):
  - Service de Pathologies infectieuses et tropicales, Hôpital Nord, CHU d'Amiens, Amiens
  - CHU ANGERS - Service des maladies infectieuses et tropicales, Angers
  - Service des Maladies infectieuses et Tropicales, Hôpital Jean Minjoz, CHU de Besançon, Besançon
  - Service de Réanimation médicale, Hôpital St André, CHU de Bordeaux, Bordeaux
  - Service de Médecine interne, Hôpital Ambroise Paré, APHP, Boulogne-Billancourt
  - Service de Cardiologie, Hôpitall Louis Pradel, Hôpitaux Est, Hospices Civils de Lyon, Bron
  - Service Maladies Infectieuses et tropicales, Hôpital Côte de Nacre, CHU de Caen, Caen
  - Service de Maladies infectieuses et tropicales, médecine interne, CH de Chambéry, Chambéry
  - Service des maladies infectieuses et tropicales, Hôpital G. Montpied, CHU de Clermont-Ferrand, Clermont-Ferrand
  - APHP Henri-Mondor - Service des maladies infectieuses et tropicales, Créteil
  - Département d'infectiologie, Complexe Bocage, Hôpital d'enfants, CHU de Dijon, Dijon
  - Service de Médecine interne polyvalente et neurologique CH de Douai, Douai
  - Service de Médecine aigue spécifique, Hôpital Raymond Poincaré, APHP, Garches
  - Service de Médecine post-urgence, infectiologie, Site de la Roche sur Yon, CHD Vendée, La Roche-sur-Yon
  - Service de Médecine infectieuse, Hôpital Nord Michallon, CHU de Grenoble, La Tronche
  - APHP BICETRE - Service des maladies infectieuses et tropicales, Le Kremlin-Bicêtre
  - Service des Maladies infectieuses et tropicales, CH Le Mans, Le Mans
  - Unité médicale d'infectiologie, Hôpital Huriez, CHU de Lille, Lille
  - Clinique de la Sauvegarde, Lyon
  - Service de Maladies infectieuses et tropicales, Hôpital Hôtel Dieu, CHU Nantes, Nantes
  - Service d'Infectiologie, Hôpital de l'Archet, CHU de Nice, Nice
  - Service des Maladies infectieuses, CH de Niort, Niort
  - Service des Maladies Infectieuses et Tropicales, Hôpital Carémeau, CHU de Nîmes, Nîmes
  - Service de Maladies infectieuses et tropicales, Hôpital de la Source, CHR Orléans, Orléans
  - APHP St Antoine, Paris
  - Service de Microbiologie, Hôpital Européen Georges Pompidou, APHP, Paris
  - Service de Maladies infectieuses et tropicales, Hôpital Necker, APHP, Paris
  - Service de Maladies infectieuses, parasitaires et tropicales, Hôpital Bichat, APHP, Paris
  - Institut Mutualiste Montsouris - Service de médecine interne, Paris
  - CH PAU - Service de Médecine interne et Maladies infectieuses, Pau
  - Service de Médecine interne, maladies infectieuses et tropicales, CHU de Poitiers, Poitiers
  - Infectiologie, médecine interne et médecine des voyages, CH d'Annecy, Pringy
  - CH QUIMPER - Service d'infectiologie, Quimper
  - Service de Médecine interne, maladies infectieuses, immunologie clinique, Hôpital R. Debré, CHU de Reims, Reims
  - Service des maladies infectieuses et réanimation médicale, Hôpital Pontchaillou, CHU de Rennes, Rennes
  - Service des Maladies infectieuses et tropicales, Hôpital Charles Nicolle, CHU de Rouen, Rouen
  - CHU St Etienne - Service des maladies infectieuses et tropicales, Saint-Priest-en-Jarez
  - Service des maladies respiratoires et infectieuses, CH de St Malo, St-Malo
  - Service des Maladies infectieuses et tropicales, Hôpital de Purpan, CHU de Toulouse, Toulouse
  - CHU Toulouse (Rangueil) Service de Cardiologie, Toulouse
  - Service Universitaire des Maladies Infectieuses et du voyageur, CH de Tourcoing, Tourcoing
  - Service de Médecine interne et maladies infectieuses, Hôpital Bretonneau, CHU de Tours, Tours
  - Service de Maladies infectieuses et tropicales, Hôpitaux de Brabois, CHU de Nancy, Vandœuvre-lès-Nancy
  - Consultation de Médecine Interne, maladies infectieuses et tropicales, CH intercommunal de Villeneuve St Georges, Villeneuve-Saint-Georges
  - Médipôle Lyon Villeurbanne, Villeurbanne

IPD SHARING:
Plan to Share IPD: Yes
There are no plans to grant public access to the full protocol, participant-level data or statistical code. Data from the RODEO trials is stored by the promotor of the trial. Data and the personal identifiers are stored separately and a special permit is required for access to the data. Data can be available on request for academic researchers when it have been analysed and published. Qualified researchers can ask for data sharing by the first author LB after the study finalization.
  Open Access This is an Open Access article distributed in accordance with the Creative Commons Attribution Non Commercial (CC BY-NC 4.0) license, which permits others to distribute, remix, adapt, build upon this work noncommercially, and license their derivative works on different terms, provided the original work is properly cited and the use is non-commercial. See: http:// creativecommons.org/licenses/by-nc/4.0/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After publication of the main manuscript

REFERENCES:
- [Derived] Lemaignen A, Bernard L, Tattevin P, Bru JP, Duval X, Hoen B, Brunet-Houdard S, Mainardi JL, Caille A; RODEO (Relais Oral Dans le traitement des Endocardites a staphylocoques ou streptOcoques) and AEPEI (Association pour l'Etude et la Prevention de l'Endocardite Infectieuse) study groups. Oral switch versus standard intravenous antibiotic therapy in left-sided endocarditis due to susceptible staphylococci, streptococci or enterococci (RODEO): a protocol for two open-label randomised controlled trials. BMJ Open. 2020 Jul 14;10(7):e033540. doi: 10.1136/bmjopen-2019-033540. PMID 32665381